CLINICAL TRIAL: NCT06523543
Title: Ultra-early Identification of Fetal Chromosomal Characteristics From Extravillous-trophoblast Cells
Acronym: CellF-Cervix
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0417
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-07

CONDITIONS: Pregnant Women
Keywords: Trophoblast cells; Endocervical canal; Fluorescent in situ hybridization (FISH); Non-invasive prenatal test; Fetal gender

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Women who are pregnant between 7 and 16 weeks of amenorrhea (WA)
  Interventions: Procedure: Inclusion (Visit 1 - Week 7-16); Diagnostic Test: Second semester of pregnancy (Visit 2 - Week 20-24); Diagnostic Test: Third semester of pregnancy (Visit 3- Week 34)

INTERVENTIONS:
Procedure: Inclusion (Visit 1 - Week 7-16) — Extraction of cervico-vaginal sampling
Diagnostic Test: Second semester of pregnancy (Visit 2 - Week 20-24) — Ultrasound examination (determination of chromosomal sex)
Diagnostic Test: Third semester of pregnancy (Visit 3- Week 34) — Ultrasound examination (determination of chromosomal sex) if this has not be done during the Visit 2 or if a new determination correcting the previous one is provided.

SUMMARY:
Demonstrate the efficacy of an ultra-early, non-invasive prenatal diagnostic method adaptable to various genetic indications to detect fetal chromosomal abnormalities.

DETAILED DESCRIPTION:
During pregnancy, biological screening for genetic diseases of the fetus cannot be implemented before the 11th week of amenorrhea whatever the technique used. This delay is long and distressing, particularly for people at high risk of transmission of genetic diseases. The presence of extravillous trophoblast cells to the cervix of the pregnant woman from the 7th week, accessible by a cervicovaginal smear non-invasive, represents new biological material representative of the fetal genome. This project aimed at evaluating the performance of a method for analyzing these trophoblast cells extra-villous at the start of pregnancy. The investigators want to evaluate performance analytical aspects of this method, that is to say, verifying that the genetic information resulting from these cells correspond to those of the fetus.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Singleton pregnancy
* Pregnancy between 7 and 16 weeks of amenorrhea (WA)
* Woman ≥ 18 years
* Woman who has signed an informed consent
* Woman affiliated to social security or equivalent scheme

Exclusions Criteria:

* Person under guardianship or curatorship
* Person placed under legal protection
* Person unable to provide the participant with informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women with a priori genetic risk
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Establish an ultra-early detection method | Visit 2 (Week 20-24)
  Collect fetal phenotypic data obtained during the second or the 3rd trimester via ultrasound echography

SECONDARY OUTCOMES:
Evaluate the ability of the method to provide a result in the context of a progressive pregnancy | Visit 2 (Week 20-24)
  * Time (minutes) elapsed between sampling and biological validation of the result
  * Number of trophoblast cells identified
  * Failure rate: number of samples for which biological signals were not successful to determine the fetal chromosomal sex
Expected benefit of ultra-early cytogenetic information | Visit 2 (Week 20-24)
  Evaluate the ability of the method to provide a rapid result and evaluate the impact of information about pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GATINOIS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France

REFERENCES:
- [Background] Bailey-Hytholt CM, Sayeed S, Kraus M, Joseph R, Shukla A, Tripathi A. A Rapid Method for Label-Free Enrichment of Rare Trophoblast Cells from Cervical Samples. Sci Rep. 2019 Aug 20;9(1):12115. doi: 10.1038/s41598-019-48346-3. PMID 31431640
- [Background] Bolnick JM, Kilburn BA, Bajpayee S, Reddy N, Jeelani R, Crone B, Simmerman N, Singh M, Diamond MP, Armant DR. Trophoblast retrieval and isolation from the cervix (TRIC) for noninvasive prenatal screening at 5 to 20 weeks of gestation. Fertil Steril. 2014 Jul;102(1):135-142.e6. doi: 10.1016/j.fertnstert.2014.04.008. Epub 2014 May 10. PMID 24825422
- [Background] Drewlo S, Armant DR. Quo vadis, trophoblast? Exploring the new ways of an old cell lineage. Placenta. 2017 Dec;60 Suppl 1(Suppl 1):S27-S31. doi: 10.1016/j.placenta.2017.04.021. Epub 2017 Apr 26. PMID 28483162
- [Background] Fritz R, Kohan-Ghadr HR, Bolnick JM, Bolnick AD, Kilburn BA, Diamond MP, Drewlo S, Armant DR. Noninvasive detection of trophoblast protein signatures linked to early pregnancy loss using trophoblast retrieval and isolation from the cervix (TRIC). Fertil Steril. 2015 Aug;104(2):339-46.e4. doi: 10.1016/j.fertnstert.2015.05.010. Epub 2015 Jun 11. PMID 26051097
- [Background] Kadam L, Jain C, Kohan-Ghadr HR, Krawetz SA, Drewlo S, Armant DR. Endocervical trophoblast for interrogating the fetal genome and assessing pregnancy health at five weeks. Eur J Med Genet. 2019 Aug;62(8):103690. doi: 10.1016/j.ejmg.2019.103690. Epub 2019 Jun 18. PMID 31226440
- [Background] Mantzaris D, Cram DS. Potential of syncytiotrophoblasts isolated from the cervical mucus for early non-invasive prenatal diagnosis: evidence of a vanishing twin. Clin Chim Acta. 2015 Jan 1;438:309-15. doi: 10.1016/j.cca.2014.09.002. Epub 2014 Sep 8. PMID 25218787
- [Background] Moser G, Drewlo S, Huppertz B, Armant DR. Trophoblast retrieval and isolation from the cervix: origins of cervical trophoblasts and their potential value for risk assessment of ongoing pregnancies. Hum Reprod Update. 2018 Jul 1;24(4):484-496. doi: 10.1093/humupd/dmy008. PMID 29608700
- [Background] Pfeifer I, Benachi A, Saker A, Bonnefont JP, Mouawia H, Broncy L, Frydman R, Brival ML, Lacour B, Dachez R, Paterlini-Brechot P. Cervical trophoblasts for non-invasive single-cell genotyping and prenatal diagnosis. Placenta. 2016 Jan;37:56-60. doi: 10.1016/j.placenta.2015.11.002. Epub 2015 Nov 11. PMID 26680636
- [Background] Shettles LB. Use of the Y chromosome in prenatal sex determination. Nature. 1971 Mar 5;230(5288):52-3. doi: 10.1038/230052b0. No abstract available. PMID 4102825